CLINICAL TRIAL: NCT04285645
Title: Efficacy of a Physiotherapy Protocol Through Preheating in the Improvement of Knee Stability and Quadriceps Strength in Rugby Players. A Randomized Clinical Study.
Brief Title: Preheating in the Improvement of Knee Stability and Quadriceps Strength in Rugby Players
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Lockdown
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Stability
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Rugby
Keywords: Rugby; Injury; Knee; Stability; Strength Training
MeSH Terms: conditions — Wounds and Injuries | interventions — Warm-Up Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session will last 15 minutes, taking place 2 days a week, over a period of 4 weeks. Prior to training, the exercise protocol will be carried out. Prior to the start of the intervention, the exercises to be performed will be explained to the participants and it will be verified that they are capable of performing them correctly.
  Interventions: Other: Warmup
- Control group (No Intervention): Athletes included in the control group will continue with their usual training routine.

INTERVENTIONS:
Other: Warmup — The intervention through exercises will consist in the application of the protocol described by Waldén et al. The objective of the application of this exercise protocol is to produce an improvement in the stability of the knee and the strength of the quadriceps. Before carrying out the exercises, a continuous race will be carried out for 5 minutes, once this first step is finished we will proceed to the realization of the exercises that will be, squats with both legs placing the hands on the hips, feet placed at the width of the shoulders, lowering with a straight back and without raising the heels of the floor, 3 series of 15 repetitions, squats on one leg with the hands on the hips and leg not supported extended forward, 3 sets of 10 repetitions with each leg and jump forward with one leg with the hands on the hips and jump back to return to the starting position, 3 sets of 10 repetitions with each leg
  Other Names: Experimental group
  Arms: Experimental group

SUMMARY:
Injuries to the lower limbs are the most common in rugby and within the lower limbs, the most common are those that affect the ligaments of the knee. That is why we will try to improve knee stability and quadriceps strength.

The aim of this study is to evaluate the effectiveness of performing a pre-workout exercise protocol to improve knee stability and quadriceps strength in rugby players.

Randomized controlled study, simple blind and with follow-up. 30 semi-professional rugby players will be randomized to the two study groups: experimental (pre-training exercise protocol that will include continuous running, squats, and squats and monopodal jumps) and control (without intervention). The intervention will last 4 weeks, with 2 weekly sessions of 15 minutes each. The study variables will be: knee stability (Y-Balance) and quadriceps strength (Single leg hop). The sample distribution will be calculated using the Kolmogorov-Smirnov test. The changes after each evaluation will be analyzed with the t-student test and with an ANOVA of repeated measures, the intra and intersubject effect will be observed. The effect size will be calculated using Cohen's formula.

It is expected to see improvement in knee stability and quadriceps strength in athletes who performed the exercise protocol, after the study period.

ELIGIBILITY:
Inclusion Criteria:

* Female rugby players
* With an age range of 18 to 30 years
* That participate in the Valencian territorial category 1
* Without diagnosis of lower limb injury at the time of starting the study

Exclusion Criteria:

* Players who suffer an injury or illness that prevents them from performing the protocol
* Are performing another specific physiotherapy program of knee stability and quadriceps strength
* Who had undergone the anterior cruciate ligament less than a year ago
* Have not signed the informed consent.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline knee stability after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done using the Y-Balance test. The barefoot sportswoman will be placed with the toes in the center of the Y marked on the floor with adhesive tape. Each of them will have six trials with each foot in each direction (anterior, posterolateral and posteromedial). Subsequently, they will have three attempts with each leg in each direction, taking the best mark of each leg in each direction. The athlete must return to the initial position without losing balance, because if she does not succeed, that attempt will be void. The distance to be measured includes from the central mark where we place the toes to the point where the patient supports the tip of the toes. The unit of measure of this measuring instrument is the centimeter. A higher score indicates greater knee stability.

SECONDARY OUTCOMES:
Change from baseline quadriceps strength after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done by applying the Single leg hop test. With this test, the quadriceps strength will be measured. With the patient in monopodal and barefoot support, and with the toes placed on a mark made on the floor with adhesive tape, he will make a leap forward, maintaining the balance at least one second. Each player will perform 6 warm-up jumps with each leg. Subsequently you will have three attempts with each leg and the greatest distance achieved with each one will be taken. The distance will be measured from the initial mark, to where the subject's heel lands, with cm being the unit of measure for the test. A greater distance indicates a greater force of quadriceps.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain